CLINICAL TRIAL: NCT04462588
Title: Are the Changes in Immature Granulocyte Count and Percentage Significant in the Decision to Continue Medical Treatment of Uncomplicated Acute Appendicitis Cases
Brief Title: Immature Granulocyte [IG] Count and Percentage for Medical Treatment of Uncomplicated Acute Appendicitis
Acronym: [IG]
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Mehmet Buğra Bozan, Professor, Assistant, Kahramanmaras Sutcu Imam University
Other Study IDs: 179
Record Dates: First submitted 2020-06-27; First posted 2020-07-08 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Acute Appendicitis Without Peritonitis; Medical Emergencies
Keywords: Uncomplicated Acute Appendisitis; Alvarado Scoring System; Immature Granulocyte Count; Immature Granulocyte Percentage
MeSH Terms: interventions — Ciprofloxacin; Injections; Appendectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical Treatment Group: Medical treatment group of uncomplicated acute appendisitis
  Interventions: Drug: Cipro 400 MG in 200 ML Injection; Drug: Flagyl I.V. RTU
- Surgery: Operated group of uncomplicated acute appendisitis
  Interventions: Procedure: appendectomy (open or laparascopic)

INTERVENTIONS:
Drug: Cipro 400 MG in 200 ML Injection — medical tratment group
  Other Names: Medical treatment of acute appendicitis
  Groups: Medical Treatment Group
Drug: Flagyl I.V. RTU — medical tratment group
  Other Names: Medical treatment of acute appendicitis
  Groups: Medical Treatment Group
Procedure: appendectomy (open or laparascopic) — appendectomy (open or laparascopic)
  Other Names: Appendectomy
  Groups: Surgery

SUMMARY:
After appendectomy was first described by Mcburney in 1889, it has been the most practiced emergency surgery in the world with the lifetime incidence of acute appendicitis being 5%-25%. Most cases are uncomplicated cases without any complications and perforation (20%-30%). Although appendectomy is still a curative therapy, medical treatment has come to the fore in uncomplicated cases after improvements in imaging methods for diagnosing acute appendicitis and especially the developments in antibiotherapy.

Medical treatment for acute appendicitis is, in fact, not a new condition. Practicing the option of elective surgery following intravenous antibiotherapy for plastron appendicitis that is among the complicated acute appendicitis has lead to further consideration of medical treatment. A number of studies conducted for this purpose suggest that conservative treatment in uncomplicated acute appendicitis may be a first-line treatment. Medical treatment of the uncomplicated acute appendicitis prevents negative appendectomies, which indicates that surgical removal of non-inflamed appendix ranging from 6% to 20%. In addition to preventing unnecessary organ loss, it ensures eliminating postoperative complications such as intestinal obstruction and wound site complications due to surgery.

Immature granulocytes (IG) are monitored in peripheral blood as immature polymorphonuclear cells because of the activation of bone marrow. Although their counts can be determined through direct inspection, they can be provided with automated systems within complete blood count parameters as well as technological developments. The increase in their number specifically suggests the activation of the bone marrow and can provide information about the infectious process before leukocytosis is observed.

This study aimed to determine the importance of IG count and percentage to evaluate the role of medical treatment and control its success in cases of uncomplicated acute appendicitis.

DETAILED DESCRIPTION:
After approval of local ethics committee (KSU Bioethics Committee, for the study with protocol number 179; dated June 19, 2019; session no. 2019/11; and decision no.: 4), the investigator's study was organized as a 1-year prospective randomized study. As a criterion for terminating the study, the expiration of 1 year or reaching the total number of patients obtained through power analysis. In the primary study endpoint, to detect a 20% difference with α = 5% and ß = 20%, a total sample size of 64 patients was reported to be necessary for achieving statistical significance.

Patients with the diagnosis of acute appendicitis over the age of 18 and treated by the same surgical team were prospectively registered to Kahramanmaraş Sütçü Imam University General Surgery Clinic between July 2019 and April 2020. Acute appendicitis was diagnosed with history, physical examination results, laboratory results, and imaging methods (Ultrasonography or Computed Tomography (CT)). As per these results, patients with Alvarado Score 7 and above were diagnosed with acute appendicitis. Patients diagnosed with complicated acute appendicitis based on imaging methods (such as perforation, periappendicular abscess formation, and plastron formation), patients who are pregnant, patients who did not want to be included were excluded from the study. Patients were informed that there were medical treatment and surgical treatment options in uncomplicated acute appendicitis and written consent was obtained from patients. For randomization purposes, patients were given balls to draw. Using this ball drawing, patients were divided into two groups as those that would receive random medical treatment (Group M) and those that would undergo direct appendectomy (Group A) (Open appendectomy or laparoscopic appendectomy). Group M was divided into two subgroups as those who responded to medical treatment within 24 h of follow-up and those who failed medical treatment. The study was terminated as the total number of 64 patients was reached because of power analysis.

In Group A, after examining the patient in the emergency, the patient was urgently taken to operation to perform appendectomy (open or laparoscopic). A complete blood count and CRP were studied on patients within the first 24 h of the postoperative course. In Group M, oral intake was discontinued on admission of patients to the clinic and intravenous ciprofloxacin (200 mg; twice a day) and metronidazole (500 mg; three times a day), which were effective for both gram-positive and gram-negative bacteria and anaerobes, were started with fluid replacement. When the duration of nonsurgical follow-up is between 12 and 24 h, there is no increase in the perforation risk. Considerable complications can be encountered after 48 h (wound site infections, wound decomposition, and other complications). Therefore, because of increased risk of perforation and the likelihood of complications as a result, the response protocol for medical treatment was restricted to 24 h. During follow-up, vital signs of patients were verified every 6 h. At the 24th h of follow-up, the patients were asked for their complaints and physical examinations were performed. Control of complete blood count, CRP, and abdominal US were performed. At the 24th hour of the follow-up, Alvarado score was repeated to patients. Patients who had no regression in the clinic and laboratory results (with an Alvarado score ≥ 7 and who had an appendix unresponsive to medical treatment according to imaging methods (with no change in diameter or increased or developed complications) were considered to be unresponsive to conservative treatment and rescue appendectomy was performed. Patients with a regression in physical examination and laboratory results (with calculating Alvarado score <7) and those with an appendix that responded to medical treatment as per imaging methods (with reduced diameter or not monitored with US) were considered to have responded to conservative treatment; and oral intake was initiated without surgery. . They were discharged from the hospital with a prescription of 1-week oral antibiotic regimen (a combination of oral ciprofloxacin 500 mg and oral metronidazole 500 mg two times daily (morning and evening)). At the end of antibiotic therapy, patients were called for control.

WBC count, neutrophil count, lymphocyte count, IG count and IG% were measured using an automated hematological analyzer (XN 3000; Sysmex Corp., Kobe, Japan) and CRP levels were measured using an automated biochemical analyzer (Cobas C-702 module, Roche Diagnostics, Basel, Sweden) from blood samples obtained at the initial admission to the emergency department and the 24th hour of the follow-up. Neutrophil to lymphocyte ratio (NLR) levels were manually calculated. The IG fraction includes promyelocytes, myelocytes, and metamyelocytes but not band neutrophils or myeloblasts. Moreover, DNI (IG percentage-%) is the IG count to white blood cell ratio.

Statistical Evaluation: IBM Statistical Package for Social Sciences for windows, Version 20.0 software package (IBM Corp., Armonk, NY, USA) was used to evaluate statistical data. Therefore, 64 patients were required to achieve 80% power to detect a difference of 10% among IG count and percentage, the means using student t-test and repeated measures ANOVA at the 0. 05 significance level.

Kolmogorov-Smirnov test was performed for the suitability of patients for normal distribution. Based on their suitability for normal distribution, paired sample t test was used to evaluate intra-group measurements in numerical data, while student t-test and Mann-Whitney U test were used in inter-group evaluation. Repeated measurement ANOVA and Scheffe's post-hoc test were used to evaluate the relationship between subgroups and appendectomy group. Note that Chi square test and Fischer's exact test were used to evaluate the categorical data. Numerical data were given as median (minimum - maximum), and categorical data were indicated in numbers (n) and percentages (%). Statistically, p<0.05 values were considered to be significant.

ELIGIBILITY:
Inclusion Criteria:

Clinically diagnosed uncomplicated acute appendisitis cases Uncomplicated acute appendicitis cases who accepted the study protocol Successfully medical treated acute appendicitis Operated uncomplicated acute appendicitis cases -

Exclusion Criteria:

Clinically diagnosed complicated acute appendisitis cases Uncomplicated acute appendicitis cases who do not accept the study protocol Patients with any type of malignancy (appendix or other organ) Patients with rheumatologic disease or blood diseases

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Elder than 18 years old
Study Population: Uncomplicated acute appendicitis cases
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Medical treatment success | Started with administration to the clinic and finished with the 24th hour of the follow up
  Defining medical treatment success with immature granulocyte count (/mm3) comparing with appendectomy group's samples
Medical treatment success | Started with administration to the clinic and finished with the 24th hour of the follow up
  Defining medical treatment success with immature granulocyte percentage (immature granulocyte count/total white blood cell count x100) comparing with appendectomy group's samples

SECONDARY OUTCOMES:
Medical treatment continue | Started with administration to the clinic and finished with the 24th hour of the follow up
  Defining medical treatment success with immature granulocyte count (/mm3) comparing with appendectomy group's samples
Medical treatment continue | Started with administration to the clinic and finished with the 24th hour of the follow up
  Defining medical treatment success with immature granulocyte percentage (immature granulocyte count/total white blood cell count x100) comparing with appendectomy group's samples
Medical treatment continue | ALVARADO Score in the first administration to the clinic and the 24th hour of the follow up
  Defining medical treatment success with ALVARADO Score comparing with appendectomy group's samples for continuing the medical treatment options

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirkil C, Yigit MV, Aygen E. Long-term results of nonoperative treatment for uncomplicated acute appendicitis. Turk J Gastroenterol. 2014 Aug;25(4):393-7. doi: 10.5152/tjg.2014.7192. PMID 25254521
- [Background] Okus A, Ay S, Karahan O, Eryilmaz MA, Sevinc B, Aksoy N. Monitoring C-reactive protein levels during medical management of acute appendicitis to predict the need for surgery. Surg Today. 2015 Apr;45(4):451-6. doi: 10.1007/s00595-014-1099-6. Epub 2014 Dec 27. PMID 25542081
- [Background] Unal Y. A new and early marker in the diagnosis of acute complicated appendicitis: immature granulocytes. Ulus Travma Acil Cerrahi Derg. 2018 Sep;24(5):434-439. doi: 10.5505/tjtes.2018.91661. PMID 30394497
- [Background] Salminen P, Tuominen R, Paajanen H, Rautio T, Nordstrom P, Aarnio M, Rantanen T, Hurme S, Mecklin JP, Sand J, Virtanen J, Jartti A, Gronroos JM. Five-Year Follow-up of Antibiotic Therapy for Uncomplicated Acute Appendicitis in the APPAC Randomized Clinical Trial. JAMA. 2018 Sep 25;320(12):1259-1265. doi: 10.1001/jama.2018.13201. PMID 30264120
- [Background] Becker P, Fichtner-Feigl S, Schilling D. Clinical Management of Appendicitis. Visc Med. 2018 Dec;34(6):453-458. doi: 10.1159/000494883. Epub 2018 Nov 24. PMID 30675493
- [Background] Wojciechowicz KH, Hoffkamp HJ, van Hulst RA. Conservative treatment of acute appendicitis: an overview. Int Marit Health. 2010;62(4):265-72. PMID 21348022
- [Background] Coccolini F, Fugazzola P, Sartelli M, Cicuttin E, Sibilla MG, Leandro G, De' Angelis GL, Gaiani F, Di Mario F, Tomasoni M, Catena F, Ansaloni L. Conservative treatment of acute appendicitis. Acta Biomed. 2018 Dec 17;89(9-S):119-134. doi: 10.23750/abm.v89i9-S.7905. PMID 30561405
- [Background] Karon BS, Tolan NV, Wockenfus AM, Block DR, Baumann NA, Bryant SC, Clements CM. Evaluation of lactate, white blood cell count, neutrophil count, procalcitonin and immature granulocyte count as biomarkers for sepsis in emergency department patients. Clin Biochem. 2017 Nov;50(16-17):956-958. doi: 10.1016/j.clinbiochem.2017.05.014. Epub 2017 May 25. PMID 28552399
- [Background] Nahm CH, Choi JW, Lee J. Delta neutrophil index in automated immature granulocyte counts for assessing disease severity of patients with sepsis. Ann Clin Lab Sci. 2008 Summer;38(3):241-6. PMID 18715852
- [Background] Unal Y, Barlas AM. Role of increased immature granulocyte percentage in the early prediction of acute necrotizing pancreatitis. Ulus Travma Acil Cerrahi Derg. 2019 Mar;25(2):177-182. doi: 10.14744/tjtes.2019.70679. PMID 30892679
- [Background] Park JS, Kim JS, Kim YJ, Kim WY. Utility of the immature granulocyte percentage for diagnosing acute appendicitis among clinically suspected appendicitis in adult. J Clin Lab Anal. 2018 Sep;32(7):e22458. doi: 10.1002/jcla.22458. Epub 2018 Apr 30. PMID 29708633
- [Background] Kirkil C, Karabulut K, Aygen E, Ilhan YS, Yur M, Binnetoglu K, Bulbuller N. Appendicitis scores may be useful in reducing the costs of treatment for right lower quadrant pain. Ulus Travma Acil Cerrahi Derg. 2013 Jan;19(1):13-9. doi: 10.5505/tjtes.2013.88714. PMID 23588973